CLINICAL TRIAL: NCT02207452
Title: A Randomized, Methodology Study to Investigate the Use of 3He-MRI Lung Ventilation and Proton MRI Perfusion Imaging to Detect Changes in Ventilation Perfusion Relationships in Chronic Obstructive Pulmonary Disease (COPD) Patients; a Proof of Concept Study.
Brief Title: Helium-3 MRI Imaging Study in COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 111175
Record Dates: First submitted 2012-01-12; First posted 2014-08-04 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Hyperpolarised helium-3; Lung Imaging; Magnetic Resonance Imaging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

ARMS (2):
- Salbutamol + Ipratropium (Other): Treatment period 1: Salbutamol 5mg nebulised, single Dose. Treatment period 2: Ipratropium 500mcg nebulised, single dose.
  Interventions: Device: He-3 MRI; Drug: Salbutamol; Drug: Ipratropium; Device: MRI
- Ipratropium + Salbutamol (Other): Treatment period 1: Ipratropium 500mcg nebulised, single dose. Treatment period 2: Salbutamol 5mg nebulised, single Dose.
  Interventions: Device: He-3 MRI; Drug: Salbutamol; Drug: Ipratropium; Device: MRI

INTERVENTIONS:
Device: He-3 MRI — Hyperpolarised helium-3 Magnetic Resonance Imaging (MRI) scan pre-bronchodilator and 1 hour post-bronchodilator (after 1 hour post-bronchodilator assessments/procedures completed).
  Other Names: Hyperpolarised Helium-3 MRI; He-3 Magnetic Resonance Imaging
Drug: Salbutamol — Salbutamol 5mg nebulised single dose
Drug: Ipratropium — Ipratropium 500mcg nebulised single dose
Device: MRI — Proton Magnetic Resonance Imaging (MRI) scan pre-bronchodilator and 1 hour post-bronchodilator (after 1 hour post-bronchodilator assessments/procedures completed).
  Other Names: 1H MRI

SUMMARY:
This protocol describes the investigation of the use of hyperpolarised helium magnetic resonance imaging (MRI) in reflecting the regional differences in lung function of moderate to severe Chronic Obstructive Pulmonary Disease (COPD) patients.

Since finalisation of the original protocol, new medications for COPD have received Market Authorisation Approvals. Protocol Amendment 02 has been prepared to include these medications in the protocol eligibility criteria and restrictions for the study.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an important cause of morbidity, mortality, and healthcare costs worldwide. COPD is characterized by progressive airflow limitation that is not fully reversible and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases. It has become clear that simple measures of airflow obstruction are inadequate to relate lung function to exercise capacity or symptoms, and that complex expressions such as dynamic hyper-inflation need to be invoked in seeking to understand overall physiology. In addition to abnormalities of air flow, gas exchange is also deranged. Therefore in considering new treatment approaches, both abnormalities need to be addressed.

Techniques to study ventilation variation and perfusion matching across the lung exist but are invasive and exacting, and do not give an indication of the anatomical distribution of changes. There is a clear need for techniques which can provide sensitive, useful and safe repeated measures reflecting regional changes in ventilation and gas exchange in COPD. This study investigates use of hyperpolarised helium magnetic resonance imaging (MRI) in reflecting the regional differences in lung function of moderate to severe COPD patients. A Beta2 bronchodilator - Salbutamol - and a anticholinergic - Ipratropium - will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of Chronic Obstructive Pulmonary Disease (COPD) diagnosis: an established clinical history of chronic pulmonary disorder in accordance with the following description by the American Thoracic Society / European Respiratory Society [ATS / ETS, 2004]

Chronic obstructive pulmonary disease is a preventable and treatable disease characterised by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and is associated with an abnormal inflammatory response of the lungs to noxious particles or gases, primarily caused by cigarette smoking. Although COPD affects the lungs, it also produces significant systemic consequences.

* The patient is clinically stable with no change in symptoms or medication, no admissions to hospital, and with neither antibiotic therapy nor systemic steroid use for at least 6 weeks prior to screening. (Screening may be rescheduled after an appropriate period of stability)
* Male and female patients aged ≥50 years
* A female patient is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) ≥40 M1U/mL and estradiol ≤ 40 pg/mL (≤140 pmol/L) is confirmatory).
* Subjects have refrained from short-acting bronchodilators for 8 hours, long-acting β2-agonists (including any long-acting β2 agonist containing inhaler) and theophyllines for 24 hours and Tiotropium, phosphodiesterase-4 (PDE4) inhibitors (e.g. Roflumilast) and ultra long-acting beta-adrenoceptor agonists (e.g. Indacaterol) for 48 hours prior to admission to the unit on study days.
* Subjects with a post-bronchodilator FEV1 to FVC ratio (FEV1/FVC) < 0.7
* Subjects with a post-bronchodilator FEV1 ≥ 30% and ≤ 80% of predicted normal for height, age and sex at screening.
* Subjects with a cigarette smoking history of ≥10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year or the equivalent). Both current and former smokers are eligible to be enrolled.
* Resting SpO2 of >90% on room air
* QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block (based on a single ECG value).
* The patient is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions, and to give informed consent.

Exclusion Criteria:

* Unstable cardiac disease or history of clinically significant arrhythmia (including established atrial fibrillation).
* Patients with a primary diagnosis of α-1 antitrypsin deficiency.
* Patients with other significant respiratory disorders.
* Patients with any acute infection, exacerbation of COPD or other unstable medical condition.
* Patients in whom inhaled beta-2 agonists or anticholinergics are contraindicated.
* Patients who have undergone thoracic surgery including lung volume reduction surgery or have conditions that prevent them from performing spirometry and other physiological testing.
* Patients who are non Magnetic Resonance Imaging (MRI) compatible (ferro-magnetic metallic implants, pacemakers) as per the MRI questionnaire.
* Patients with renal complaints relating to potential adverse reactions to Gd-DTPA intravascular MRI contrast agent.
* Patients who suffer from claustrophobia.
* The patient has participated in a clinical trial and has received an investigational product within the following time period prior to the first study day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) of that study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Subjects must abstain from taking prescription (not related to their COPD) or nonprescription drugs (including vitamins and dietary or herbal supplements), within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first study day until completion of the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-08-05 (Actual); Primary Completion 2011-07-04 (Actual); Study Completion 2011-07-04 (Actual)

PRIMARY OUTCOMES:
Changes in Oxygen Saturation | Baseline measurement at screening visit (up to 30 days prior to first dose). Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post dose), for both treatment periods.
  To correlate changes in oxygen saturation pre- and post- bronchodilator (as a reflection of ventilation/perfusion matching) with changes in distribution of regional ventilation/perfusion (V/Q) demonstrated by hyperpolarized helium ventilation MRI/spatially registered proton perfusion.
Changes in distribution of regional ventilation/perfusion assessed by spatially registered Helium-3 Magnetic Resonance Imaging (MRI) and proton perfusion MRI. | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  To correlate changes in oxygen saturation pre- and post- bronchodilator (as a reflection of ventilation/perfusion matching) with changes in distribution of regional ventilation/perfusion (V/Q) demonstrated by hyperpolarized helium ventilation MRI/spatially registered proton perfusion.

SECONDARY OUTCOMES:
Changes in lung volumes. | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  To compare lung volumes assessed by plethysmography with registered Helium-3 ventilation MRI and proton MRI.
Changes in standard lung function parameters. | Baseline measurement at screening visit (up to 30 days prior to first dose). Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post dose), for both treatment periods.
  To compare changes in ventilatory parameters as assessed by pulmonary function tests (spirometry) and Helium-3 MRI.
Number of adverse events | From screening (up to 30 days prior to Day 1) to follow-up (7-14 days after last dose).
  To monitor the safety of Helium-3 MRI through adverse events and clinical lung function.
Reproducibility of Helium-3 MRI | Pre-treatment Day 1 (0.5-2 hours pre-dose) for both treatment periods.
  To evaluate reproducibility of Helium-3 MRI (pre-bronchodilator) over a 2 week period.
Symptomatic effects of bronchodilators. | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  To correlate the symptomatic effects of bronchodilators with measures of lung function derived from physiological measures and from 3He MRI and proton MRI.
Regional lung oxygen uptake (pO2) | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  To compare regional oxygen uptake (direct V/Q) from 3He MRI pO2 mapping with regional V/Q derived from the ratio of 3He ventilation MRI (V) and spatially registered contrast enhanced proton perfusion MRI (Q).
Change in breathlessness | From screening (up to 30 days prior to Day 1) to follow-up (7-14 days after last dose).
  Change in breathlessness according to the Modified Borg Scale of breathlessness.
Helium-3 apparent diffusion coefficient measurements | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  Helium-3 apparent diffusion coefficient measurements (sensitivity to emphysematous alveolar destruction and minor airway size).
Distribution of flow velocities in major airways | Pre-treatment Day 1 (0.5-2 hours pre-dose) and post-dose Day 1 (1 hour post-dose), for both treatment periods.
  Distribution of flow velocities in major airways assessed by helium-3 MRI
Changes in dyspnoea | From screening (up to 30 days prior to first dose) to follow-up (7-14 days after last dose).
  Changes in shortness of breath/air hunger monitored throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Sheffield, United Kingdom

REFERENCES:
- See also: Results for study 111175 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111175?search=study&search_terms=111175#rs